CLINICAL TRIAL: NCT00003833
Title: The Clinical and Pathological Significance of Allelic Imbalance of 8p in Patients With Colorectal Cancer
Brief Title: Genetic Study in Patients With Stage II or Stage III Colon Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Other Study IDs: NCCTG-984654; CDR0000066990 (Registry Identifier: PDQ (Physician Data Query)); CAN-NCIC-CO9PATH
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Chromosome Mapping

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Normal and tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal and tumor tissue pairs: Matched normal and tumor DNA is analyzed for 8p allelic imbalance with at least 8 markers: D8S262 and D8S1825 localized to 8p23, D8S254 and D8S261 at 8p22, D8S560 and D8S136 at 8p21, and D8S1820 and D8S283 at 8p12. Normal/tumor tissue pairs are used for fine mapping studies.
  Interventions: Genetic: DNA stability analysis; Genetic: gene mapping

INTERVENTIONS:
Genetic: DNA stability analysis
Genetic: gene mapping

SUMMARY:
RATIONALE: Genetic studies may help in understanding the genetic processes that cause some types of cancer.

PURPOSE: Genetic trial to study certain genes of patients who have stage II or stage III colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the adverse prognostic significance of 8p allelic imbalance (AI) in patients with colon cancer.
* Determine if patient prognosis is dependent on the region of 8p AI.
* Perform fine mapping studies to further localize the putative tumor suppressor gene(s) on 8p.
* Perform multicolor FISH to examine the role that 8p loss and 8q gain play in the prognosis of patients whose tumors exhibit 8p AI.

OUTLINE: Matched normal and tumor DNA is analyzed for 8p allelic imbalance with at least 8 markers: D8S262 and D8S1825 localized to 8p23, D8S254 and D8S261 at 8p22, D8S560 and D8S136 at 8p21, and D8S1820 and D8S283 at 8p12. Normal/tumor tissue pairs are used for fine mapping studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of resectable stage II or III adenocarcinoma of the colon
* Participated in NCCTG-914653
* DNA extracted from both normal and tumor tissue

PATIENT CHARACTERISTICS:

Age

* Under 70

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced colon cancer previously participating in NCCTG-914653.
Sampling Method: Non-Probability Sample
Enrollment: 598 (Actual)
Dates: Start 1999-02; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Goldberg, MD, Study Chair — Mayo Clinic
Locations (59):
- St. Mary's/Duluth Clinic Health System, Duluth, Minnesota, United States
- Canada (58):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Lethbridge Cancer Clinic, Lethbridge, Alberta
  - Nanaimo Cancer Clinic, Nanaimo, British Columbia
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - Prostate Centre at Vancouver General Hospital, Vancouver, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - St. Paul's Hospital - Vancouver, Vancouver, British Columbia
  - G. Steinhoff Clinical Research, Victoria, British Columbia
  - Moncton Hospital, Moncton, New Brunswick
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cape Breton Cancer Centre, Sydney, Nova Scotia
  - Royal Victoria Hospital, Barrie, Barrie, Ontario
  - William Osler Health Centre, Brampton, Ontario
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Hamilton and District Urology Association, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - York County Hospital, Newmarket, Ontario
  - North York General Hospital, Ontario, North York, Ontario
  - Male Health Centre/CMX Research Inc., Oakville, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Scarborough Hospital - General Site, Scarborough Village, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Women's College Campus, Sunnybrook and Women's College Health Science Center, Toronto, Ontario
  - Saint Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Centre Hospitalier Regional de Lanaudiere, Joliette, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Kells Medical Research Group Inc., Pointe-Claire, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Hopital du Saint-Sacrament, Quebec, Québec, Quebec
  - Centre Hospitalier Regional de Rimouski, Rimouski, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Lions Gate Hospital, North Vancouver